CLINICAL TRIAL: NCT04160936
Title: The Effect of Peritubal Infiltration With Bupivacaine Around Nephrostomy Tract on Postoperative Pain Control After Percutaneous Nephrolithotomy
Brief Title: The Efficacy of Peritubal Analgesic Infiltration in Postoperative Pain Following Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saddam Al Demour (Other)
Responsible Party: Sponsor-Investigator, Saddam Al Demour, Assistant Professor, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sad2007
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group :infiltration with 0.25% bupivacaine post-op (Active Comparator): At the end of the procedure ( surgery), In the patients of the study group, the 23-gauge, 90mm spinal needle will inserted up to the renal capsule under fluoroscopic guidance along the nephrostomy tube at 6 and 12 o'clock positions (cranial and caudal); then 20 ml of 0.25% bupivacaine will infiltrated into the nephrostomy tract, while gradually withdrawing the needle from renal capsule to the skin thereby infiltrating the renal capsule, perinephric fat, muscles, subcutaneous tissue and skin
  Interventions: Drug: Marcaine Injectable Product
- control group , no anesthesia infiltration post-op (No Intervention): control group: no anesthesia infiltration had been given post opertatively

INTERVENTIONS:
Drug: Marcaine Injectable Product — Following PCNL under general anesthesia, patients will receive 0.25% Bupivacaine ( Marcaine) local anesthetic infiltration
  Other Names: Sensorcaine Injectable Product
  Arms: study group :infiltration with 0.25% bupivacaine post-op

SUMMARY:
The investigators aim to investigate the effect of peritubal local anesthetic infiltration on pain scores and analgesic consumption in patients who underwent percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
The investigators aim to investigate the effect of peritubal local anesthetic on pain scores and analgesic consumption in patients who underwent percutaneous nephrolithotomy. Patients aged between 18 and 65 years with renal stone >2 cm will be included in this study .The patients will be divided into two groups. In Group A , the drug will be infiltrated to the renal capsule, perinephric fat, muscles, subcutaneous tissue, and skin under fluoroscopy with 0.25 percent bupivacaine. This is a widely-used procedure by surgeons in the world. In Group B, no anesthetic will be infiltrated after the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* body mass index <35,
* renal stone size >2.0 cm.

Exclusion Criteria:

* patients having supra-costal puncture.
* excessive intraoperative bleeding.
* renal stones requiring more than a single puncture.
* surgical procedure extending more than 3 hours.
* urinary tract infection.
* severe cardiopulmonary disease.
* abnormal renal function tests.
* allergy to local anesthetics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS ) | 1, 4, 8, 12, 24, and 48 hours
  Visual Analogue Scale (VAS), the patient is asked to describe the level of pain on a visual scale at rest at 1, 4, 8, 12, 24, and 48 hours
Dynamic Visual Analogue Scale (DVAS) | 1 hour, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours
  Dynamic Visual Analogue Scale (DVAS), the patient is asked to describe the level of pain on a visual scale during breathing at 1, 4, 8, 12, 24, and 48 hours

SECONDARY OUTCOMES:
The time for the first opioid demand | 48 hours
  first post op time for analgesia
the number of opioid demands | 48 hours
  total number of opioid given to the patient
total opioid consumption | 48 hours
  total amount of opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Saddam AlDemour, professor, Principal Investigator — The University of Jordan
Locations (1):
- Saddam Al Demour, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
no IPD sharing plan

REFERENCES:
- [Derived] Al Demour SH, Halalsheh OM, Al-Azab RS, Al-Zubi MT, Al-Rawashdah SF, Ibrahim MM, Abubaker AK, Aloweidi AS, Almustafa MM. The efficacy of bupivacaine infiltration along nephrostomy tract on postoperative pain control and opioid consumption after PCNL: a prospective randomized controlled trial. Eur Rev Med Pharmacol Sci. 2023 Jun;27(11):4951-4959. doi: 10.26355/eurrev_202306_32612. PMID 37318469